CLINICAL TRIAL: NCT04649476
Title: A Randomized Phase II Study of Neoadjuvant PD-1 Blockade Alone or Plus TPF Induction Chemotherapy for Resectable Local Advanced Oral Squamous Cell Carcinoma
Brief Title: Neoadjuvant PD-1 Blockade in Resectable Oral Squamous Cell Carcinoma
Acronym: NEOPBOSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital of Stomatology, Wuhan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Gang Chen, Chief physician, Professor, Hospital of Stomatology, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HStomatologyWuhan
Record Dates: First submitted 2020-11-18; First posted 2020-12-02 (Actual); Results first posted 2024-04-12 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Neoadjuvant; Oral squamous cell carcinoma; PD-1 blockade; Camrelizumab; TPF induction chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — camrelizumab; Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant PD-1 blockade alone (Experimental): The participants will receive 3 doses of neoadjuvant PD-1 blockade. Then the participants will take a radical surgery followed by radiotherapy or chemoradiotherapy if necessary.
  Interventions: Drug: Camrelizumab
- Neoadjuvant PD-1 blockade plus TPF induction chemotherapy (Experimental): The participants will receive 3 doses of PD-1 blockade and 2 courses of TPF induction chemotherapy. Then the participants will take a radical surgery followed by radiotherapy or chemoradiotherapy if necessary.
  Interventions: Drug: Camrelizumanb plus TPF

INTERVENTIONS:
Drug: Camrelizumab — The participants will receive camrelizumab (200 mg) intravenous infusion each 2-week cycle for 3 cycles prior to surgery.
  Other Names: SHR-1210
  Arms: Neoadjuvant PD-1 blockade alone
Drug: Camrelizumanb plus TPF — The participants will receive camrelizumab (200 mg) through intravenous infusion each 2-week cycle, and docetaxel (T) 75 mg/m2, cisplatin (P) 75 mg/m2, 5-Fluorouracil (F) 750 mg/m2 through intravenous infusion each 3-week cycle for 2 cycles.
  Other Names: Docetaxel, Cisplatin, 5-Fluorouracil
  Arms: Neoadjuvant PD-1 blockade plus TPF induction chemotherapy

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of neoadjuvant PD-1 blockade alone or neoadjuvant PD-1 blockade plus TPF induction chemotherapy in subjects with resectable local advanced oral squamous cell carcinoma.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the safety and feasibility of neoadjuvant PD-1 blockade alone or neoadjuvant PD-1 blockade plus TPF induction chemotherapy in subjects with resectable local advanced OSCC. And on this basis, we will explore the changes of the profiles and functions of immune cells within tumors, lymph nodes and peripheral blood after the experimental interventions, as well as their correlation with the patients' response and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented oral squamous cell carcinoma (biopsy required).
2. Local advanced oral squamous cell carcinoma (clinical stage T1-2N1-3M0, T3-4aN0-3M0) with resection option for potential cure, as assessed by a faculty surgeon at Hospital of Stomatology, Wuhan University.
3. Distant metastasis is excluded by chest CT and emission computed tomograph.
4. Adequate organ function as follows: 1) Leukocyte count ≥ 2,000/mm3; 2) Absolute neutrophil count ≥ 1,000/mm3; 3) Platelet count ≥ 100,000/mm3; 4) Hemoglobin ≥ 90 g/L; 5) Serum albumin ≥30 g/L; 6) Total bilirubin ≤ 1.5 × upper limit of normal (ULN); 7) AST (SGOT) and ALT (SGPT) < 2.5 × ULN; 8) ALP ≤ 2.5 × ULN; 9) Prothrombin time-international normalized ratio ≤ 1.5; 10) Serum creatinine ≤ 1.5 × ULN; 11) INR/PT≤ 1.5; 12) TSH ≤ ULN.
5. ECOG performance status 0-1.
6. Female patient tested HCG negative in serum or urine within 7 days prior to the start of investigational product. Both patient and partner must agree to use contraception prior to study entry and for the duration of study participation and for up to 120 days after the last dose of PD-1 blockade.
7. Patient understands the study regimen, its requirements, risks and discomforts and is able and willing to sign the informed consent form.

Exclusion Criteria:

1. History of ≥ 3 grade immune related adverse events (irAEs) or have not recovered to ≤ 1 grade irAEs from previous treatment.
2. History of other treatments for cancer, including surgery, chemotherapy, radiotherapy or molecular targeted therapy within past 5 years.
3. Previous therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 or any other antibody targeting T cell co-regulatory pathways.
4. Active autoimmune disease or history of refractory autoimmune disease.
5. Active systemic infection requiring therapy.
6. Patients who are receiving psychotropic drug or alcohol/drug abuse.
7. Subjects with concurrent other active malignancies.
8. HIV or untreated active HBV or HCV infections, or vaccinated (HBV, flu, varicella, etc) within 4 weeks before recruitment.
9. Uncontrollable systemic diseases, including diabetes, hypertension, etc.
10. History of stroke or transient ischemic attack within past 6 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2024-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, MD, Principal Investigator — Hospital of Stomatology, Wuhan University
Locations (1):
- Hospital of Stomatology, Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu YT, Liu HM, Ren JG, Zhang W, Wang XX, Yu ZL, Fu QY, Xiong XP, Jia J, Liu B, Chen G. Immune-featured stromal niches associate with response to neoadjuvant immunotherapy in oral squamous cell carcinoma. Cell Rep Med. 2025 Mar 18;6(3):102024. doi: 10.1016/j.xcrm.2025.102024. PMID 40107247
- [Derived] Liu HM, Xiong XP, Yu ZL, Shao Z, Chen GL, Liu YT, Wang XX, Fu QY, Cheng XX, Li J, Zhang JL, Li B, Gong HY, Zhong YH, Zhang W, Jia J, Liu B, Chen G. Neoadjuvant immunotherapy with or without chemotherapy in locally advanced oral squamous cell carcinoma: Randomized, two-arm, phase 2 trial. Cell Rep Med. 2025 Feb 18;6(2):101930. doi: 10.1016/j.xcrm.2025.101930. Epub 2025 Jan 30. PMID 39889711

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant PD-1 Blockade Alone | Neoadjuvant PD-1 Blockade Plus TPF Induction Chemotherapy
Started | 34 | 34
Completed | 34 | 32
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neoadjuvant PD-1 Blockade Alone | Neoadjuvant PD-1 Blockade Plus TPF Induction Chemotherapy | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 29 | 57
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.4) | 49.5 (10.0) | 50.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 28 | 31 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 34 | 34 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 34 | 34 | 68
Tumor site [Count of Participants; unit: Participants]
  Oral tongue | 18 | 18 | 36
  Gingiva | 5 | 3 | 8
  Floor of mouth | 4 | 4 | 8
  Buccal mucosa | 7 | 9 | 16
Smoking history [Count of Participants; unit: Participants]
  Current or former | 24 | 22 | 46
  Never | 10 | 12 | 22
Alcohol use history [Count of Participants; unit: Participants]
  Current or former | 15 | 18 | 33
  Never | 19 | 16 | 35
Clinical T-stage [Count of Participants; unit: Participants] — Classification of patients of oral squamous cell carcinoma based on T stage
  Participants
    T2 (Tumour more than 2 cm but not more than 4 cm in greatest dimension) better outcomes | 6 | 9 | 15
    T3 (Tumour more than 4 cm in greatest dimension) | 19 | 18 | 37
    T4a (Tumour invades through cortical bone, maxillary sinus) worse outcomes | 9 | 7 | 16
Clinical N-stage [Count of Participants; unit: Participants] — Classification of patients of oral squamous cell carcinoma based on N stage
  Participants
    N0 (No regional lymph node metastasis) better outcomes | 23 | 13 | 36
    N1 (Metastasis in a single ipsilateral lymph node, 3 cm or less in great est dimension) | 6 | 10 | 16
    N2 (Lymph node metastasis more than 3 cm but no more than 6 cm in greatest dimension) worse outcomes | 5 | 11 | 16
PD-L1 combined positive score [Count of Participants; unit: Participants] — The expression of programmed cell death-ligand 1 (PD-L1) in patients was carried out using immunohistochemical staining. Combined positive score (CPS) of PD-L1 was defined as the total number of PD-L1-stained cells (including tumor cells, tumor-associated lymphocytes, and macrophages) divided by the total number of viable tumor cells, multiplied by 100. The range was from 0-100. PD-L1>1 was considered as cut-off value for derermine positive expression of PD-L1 in oral squamous cell carcinoma.
  Participants
    <1 (Considered as negative PD-L1 expression) worse outcomes | 16 | 13 | 29
    1-19 (Considered as positive PD-L1 expression) | 12 | 18 | 30
    >=20 (Considered as positive PD-L1 expression) better outcomes | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response.
Description: Pathologic response of resected tumors and lymph nodes to neoadjuvant PD-1 blockade alone or neoadjuvant PD-1 blockade plus TPF induction chemotherapy. Hematoxylin and eosin (H&E)-stained slides of entire tumor and all sampled lymph nodes were scanned and assessed by two independent pathologists. The entire tumor bed and all sampled lymph nodes were examined histologically in patients who had pathological complete response (pCR), which was defined as the absence of viable tumor in all slides. MPR was defined as the presence of 10% or less viable residual tumor in the resected tumor specimens. Pathological partial response (pPR) was defined as presence of more than 10% and less than 50% viable residual tumor and pathological non-response (pNR) was defined as presence of more than 50% viable residual tumor in the resected tumor specimens. Pathologic response was defined as sum of pCR and MPR.
Time Frame: 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant PD-1 Blockade Alone | Neoadjuvant PD-1 Blockade Plus TPF Induction Chemotherapy
Number analyzed (Participants) | 34 | 34
Participants
  Number of participants who had no response | 25 | 2
  Number of participants who had partial response | 4 | 4
  Number of Participants Pathologic response (pCR+MPR) | 5 | 26
  Non-evaluable | 0 | 2

2. Secondary Outcome: Radiographic Response.
Description: Radiographic response of tumors and lymph nodes to neoadjuvant PD-1 blockade alone or neoadjuvant PD-1 blockade plus TPF induction chemotherapy were evaluated by enhanced computed tomography examinations and defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Complete Response (CR) was defined as disappearance of all target lesions. Partial Response (PR) was defined as >=30% decrease in the sum of the longest diameter of target lesions. Stable disease (SD) was defined as <20% increase and <30% decrease in the sum of the longest diameter of target lesions. Progressive disease (PD) was defined as >=20% increase in the sum of the longest diameter of target lesions. Overall Response (OR) = CR + PR.
Time Frame: 8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant PD-1 Blockade Alone | Neoadjuvant PD-1 Blockade Plus TPF Induction Chemotherapy
Number analyzed (Participants) | 34 | 34
Participants
  CR (Complete response) | 0 | 0
  PR (Partial response) | 3 | 16
  SD (Stable disease) | 20 | 14
  PD (Progressive disease) | 11 | 1
  Non-evaluable | 0 | 3

3. Secondary Outcome: Event-free Survival (EFS) Rate on Each Treatment Arm.
Description: EFS is the time from the date of randomization to the date of first record of disease progression as defined by RECIST 1.1.
Time Frame: 24 months.
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS) on Each Treatment Arm.
Description: OS is the time from randomization to death due to any cause.
Time Frame: 24 months.
Reporting Status: Not Posted

5. Secondary Outcome: Adverse Events (AEs).
Description: Number of participants experiencing any sign, symptom, disease, or worsening of preexisting conditions temporally associated with the experimental interventions or irrespective of the experimental interventions.
Time Frame: 24 months.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Changes in the Level of Circualting Exosomal PD-L1.
Description: The level of circulating exosomal PD-L1 at serial time points pre- and on-treatment, as detected by enzyme-linked immunosorbent assay (ELISA).
Time Frame: 24 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The specific period of time over which adverse events were collected is initiated from the begining of neoadjuvant treatment and end up with the adjuvant radiotherapy after surgery, up to 4 months
Arm/Group | Neoadjuvant PD-1 Blockade Alone | Neoadjuvant PD-1 Blockade Plus TPF Induction Chemotherapy
All-Cause Mortality (participants affected / at risk) | 0/34 | 1/34
Serious Adverse Events (participants affected / at risk) | 2/34 | 11/34
Other Adverse Events (participants affected / at risk) | 34/34 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant PD-1 Blockade Alone (N=34) | Neoadjuvant PD-1 Blockade Plus TPF Induction Chemotherapy (N=34)
Alanine aminotransferase increased (Hepatobiliary disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 10 (10)
White blood cell decreased (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Creatine kinase increased (Cardiac disorders) | 1 (1) | 0 (0)
Creatinine increased (Renal and urinary disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant PD-1 Blockade Alone (N=34) | Neoadjuvant PD-1 Blockade Plus TPF Induction Chemotherapy (N=34)
Reactive cutaneous capillary endothelial proliferation, RCCEP (Skin and subcutaneous tissue disorders) | 29 (29) | 24 (24)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 25 (25)
Mucositis oral (Skin and subcutaneous tissue disorders) | 6 (6) | 8 (8)
Creatinine increased (Renal and urinary disorders) | 6 (6) | 15 (15)
GGT increased (Hepatobiliary disorders) | 4 (4) | 5 (5)
Vomiting (Gastrointestinal disorders) | 0 (0) | 10 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 28 (28)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 5 (5) | 13 (13)
Platelet count decreased (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Blood lactate dehydrogenase increased (Hepatobiliary disorders) | 2 (2) | 9 (9)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
ALT increased (Hepatobiliary disorders) | 4 (4) | 11 (11)
AST increased (Hepatobiliary disorders) | 2 (2) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 10 (10)
Creatine kinase increased (Cardiac disorders) | 0 (0) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-03-25): https://cdn.clinicaltrials.gov/large-docs/76/NCT04649476/Prot_SAP_ICF_000.pdf